CLINICAL TRIAL: NCT02710877
Title: Pain Management During Labor: Use of Intermittent Drug Delivery Devices for Obstetric and Neonatal Outcome Improvement and Health-care Burden Reduction
Brief Title: Intermittent Automated Devices for Labor Analgesia in Emilia Romagna
Acronym: PA-RER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped funding by Regional Healthcare System.
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Laura Rinaldi, Medical Doctor, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 274/13
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Labor Pain
Keywords: epidural analgesia; patient controlled analgesia; obstetric outcome
MeSH Terms: conditions — Labor Pain | interventions — Levobupivacaine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Programmed Intermittent bolus (PIEB) (Experimental): Intervention: epidural analgesia through administration of a mixture of levobupivacaine 0,0625% and sufentanil 4 mcg. Intermittent bolus of 10 ml mixture every 75 minutes. Patient controlled bolus of 5 ml same mixture, lock-out 15 minutes.
  Interventions: Device: Programmed Intermittent bolus; Drug: Levobupivacaine; Drug: Sufentanil 4 mcg
- Manuale epidural bolus (TOP-UP) (Active Comparator): Intervention: manual epidural bolus of 15 ml levobupivacaine 0,0625% and sufentanil 5 mcg on maternal request.
  Interventions: Other: Manual epidural bolus; Drug: Levobupivacaine; Drug: Sufentanil 5 mcg

INTERVENTIONS:
Device: Programmed Intermittent bolus — Programmed epidural bolus of 10 ml mixture every 75 minutes, plus patient controlled bolus of 5 ml same mixture; lock-out 15 minutes.
  Other Names: PIEB
  Arms: Programmed Intermittent bolus (PIEB)
Other: Manual epidural bolus — Epidural bolus of 15 ml levobupivacaine and sufentanyl 10 mcg or 5 mcg administered by anesthesist on maternal request.
  Other Names: TOP-UP
  Arms: Manuale epidural bolus (TOP-UP)
Drug: Levobupivacaine — Levobupivacaine 0,0625% through peridural catheter
  Other Names: CHIROCAINE
Drug: Sufentanil 4 mcg — Sufentanil 0,4 mcg/ml through peridural catheter
  Other Names: FENTATIENIL
  Arms: Programmed Intermittent bolus (PIEB)
Drug: Sufentanil 5 mcg — Sufentanil 5 mcg through peridural catheter
  Other Names: FENTATIENIL
  Arms: Manuale epidural bolus (TOP-UP)

SUMMARY:
The study aims to determine whether the use of automated intermittent devices for labor analgesia could prevent the increase of instrumental deliveries, with same analgesia.

Moreover it will evaluate if automated devices can allow a reduction of health-care burden.

DETAILED DESCRIPTION:
Epidural analgesia is recognized as the most effective technique to control labor pain, although its possible adverse events. Continuous epidural administration of local anesthetics can stabilize the analgesic block and reduce the anesthesiologists' workload but is associated with an increase in operative vaginal delivery.

Epidural intermittent boluses performed by anesthetist are associated to reduction of dosages, but they could provide insufficient analgesia and they involve the constant anesthetist's presence in the operating room.

This is a multicenter randomized controlled trial with two arms, funded by grant of Regione Emilia Romagna, in which we will compare two different epidural analgesia protocols: anesthesiologist's supervised versus intermittent boluses with PCEA.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women at full-term pregnancy single fetus and vertex presentation, hospitalized for harbingers of labor and cervical dilation less than 5 cm
2. Numeric Rate Scale > 5

Exclusion Criteria:

1. patients aged under 18 years
2. patients with ongoing administration of oxytocin
3. patients with no indications to epidural analgesia
4. patients with inability to place the epidural catheter for technical difficulty
5. patients with parenteral administration of opioids
6. multiparous women
7. patients unable to understand the objectives and procedures of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2014-12-23 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of instrumental delivery | Through labor completion
  Vaginal delivery obtained through vacuum device intervention decided independently by the obstetrician on duty, according to defined local protocols and according to the conditions of the mother and fetus.

SECONDARY OUTCOMES:
Adequate analgesia | Labor length since peridural catheter insertion until delivery
  Mean Numeric Rate Scale values < 5 through labor analgesia
Total amount of local anesthetic | Labor length since peridural catheter insertion until delivery
  Total amount of levobupivacaine (mg)
Time-related amount of local anesthetic | Labor length since peridural catheter insertion until delivery
  Amount of levobupivacaine for minute of analgesia (mg/min)
Motor block episodes | Labor length since peridural catheter insertion until delivery
  Number of patients with motor block episodes, defined by modified Bromage score >1
Anesthesiologist working time | Labor length since peridural catheter insertion until delivery
  Total time spent in labor room by anesthesiologist (minutes)
Health economic assessment | Labor length since peridural catheter insertion until delivery
  Total epidural analgesia charge

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Girardis, PhD, Study Director — University of Modena and Reggio Emilia
Locations (3):
- Italy (3):
  - Ospedale Ramazzini di Carpi, Carpi, MO
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists Committee on Obstetric Practice. ACOG committee opinion. No. 339: Analgesia and cesarean delivery rates. Obstet Gynecol. 2006 Jun;107(6):1487-8. doi: 10.1097/00006250-200606000-00060. PMID 16738188
- [Background] Anim-Somuah M, Smyth RM, Jones L. Epidural versus non-epidural or no analgesia in labour. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD000331. doi: 10.1002/14651858.CD000331.pub3. PMID 22161362
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Liu EH, Sia AT. Rates of caesarean section and instrumental vaginal delivery in nulliparous women after low concentration epidural infusions or opioid analgesia: systematic review. BMJ. 2004 Jun 12;328(7453):1410. doi: 10.1136/bmj.38097.590810.7C. Epub 2004 May 28. PMID 15169744
- [Background] Benedetto C, Marozio L, Prandi G, Roccia A, Blefari S, Fabris C. Short-term maternal and neonatal outcomes by mode of delivery. A case-controlled study. Eur J Obstet Gynecol Reprod Biol. 2007 Nov;135(1):35-40. doi: 10.1016/j.ejogrb.2006.10.024. Epub 2006 Nov 28. PMID 17126475
- [Background] Capogna G, Camorcia M, Stirparo S, Farcomeni A. Programmed intermittent epidural bolus versus continuous epidural infusion for labor analgesia: the effects on maternal motor function and labor outcome. A randomized double-blind study in nulliparous women. Anesth Analg. 2011 Oct;113(4):826-31. doi: 10.1213/ANE.0b013e31822827b8. Epub 2011 Jul 25. PMID 21788309
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Usha Kiran TS, Thakur MB, Bethel JA, Bhal PS, Collis RE. Comparison of continuous infusion versus midwife administered top-ups of epidural bupivacaine for labour analgesia: effect on second stage of labour and mode of delivery. Int J Obstet Anesth. 2003 Jan;12(1):9-11. doi: 10.1016/s0959-289x(02)00158-9. PMID 15676314